CLINICAL TRIAL: NCT03880799
Title: The MEDITATE-BC Study: Mindfulness-Enhanced Decision Intervention To Aid Treatment Election - Breast Cancer
Acronym: MEDITATE-BC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Katharine Yao, MD, Chief, Division of Surgical Oncology, Endeavor Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EH18-203
Record Dates: First submitted 2018-11-27; First posted 2019-03-19 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer; Surgery
Keywords: Mindfulness; Surgical Decision Making
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: non-randomized feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Intervention (Experimental): Newly diagnosed breast cancer patients who undergo a mindfulness session before their surgical appointment.
  Interventions: Behavioral: Mindfulness Session

INTERVENTIONS:
Behavioral: Mindfulness Session — one hour mindfulness session conducted by a certified mindfulness teacher with the breast cancer patient

SUMMARY:
In this study the investigators propose to pilot test a brief, mindfulness shared decision making intervention that begins shortly after receiving a diagnosis of breast cancer. A mindfulness instructor will conduct an hour long session with consented participants before the scheduled surgical appointment. The investigators hypothesize that a mindfulness intervention delivered shortly after receiving a diagnosis of breast cancer may ultimately lead to increased decisional satisfaction and alignment to participant's values and preferences, and decreased anxiety. To measure this endpoint, participants will complete three surveys via REDCap- at baseline, before surgery, and 6 months postoperatively. Surveys will include questions on quality of life, anxiety, and participant satisfaction with the mindfulness program.

DETAILED DESCRIPTION:
The primary aim of this study is to identify if a mindfulness intervention is feasible before the participant has their surgical consultation. The secondary aim is to measure the impact of the mindfulness intervention on participant reported outcomes including anxiety, quality of life and decisional satisfaction. Newly diagnosed female breast cancer patients will be contacted over the phone after the patient learns of their diagnosis but prior to their surgical appointment to discuss surgical options. Verbal consent will be obtained over the phone and the participant will be directed to complete an online survey to answer baseline questions on their anxiety and quality of life as well as to provide their contact information and availability in order to schedule a mindfulness session with a certified mindfulness teacher. The participant will then proceed to an hour-long mindfulness exercise geared to help women apply these techniques to the decisional making process. The goal is to empower women to approach their diagnosis and treatment decisions with greater stability and improve their ability to focus on their values and preferences instead of just focusing on the diagnosis. This will be measured by administering patient reported outcomes (PROs) via REDCap online surveys at three timepoints. The first PRO "baseline survey" is administered after the participant enrolls but before the mindfulness session. The second PRO "before surgery survey" is completed after the surgical consultation but prior to the scheduled surgery. The final PRO "6-month survey" is administered 6 months after the surgery to measure quality of life, anxiety, and participant satisfaction with the mindfulness program. The investigators hypothesize that a mindfulness intervention delivered shortly after receiving a diagnosis of breast cancer may ultimately lead to increased decisional satisfaction and alignment to participant's values and preferences, and decreased anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Females >20 and < 70 years of age
2. History of contralateral breast cancer in the past is acceptable
3. Patients seeking second opinion for diagnosis are eligible
4. Clinical AJCC stage 0-III breast cancer
5. Patients who have an in breast tumor recurrence are eligible
6. English Speaking
7. Willing to fill out surveys required for the study
8. Gene mutation carriers are eligible
9. Neoadjuvant therapy patients are eligible

Exclusion Criteria:

1. AJCC Stage IV breast cancer
2. Unwilling to fill out surveys for the study
3. Patients with a distant recurrence
4. Patients unaware of their diagnosis

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2020-02-08 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Acceptability of a mindfulness intervention prior to the surgical consultation measured by adherence to the intervention. | 1 year
  The number of patients who have successfully completed their mindfulness session with the mindfulness instructor. Zero being not one completion, twenty-five being all have completed the mindfulness session.
Acceptability of a mindfulness intervention following the surgical consultation measured by adherence to the follow up session. | 1 year
  The number of patients who have successfully completed their mindfulness follow up session with the mindfulness instructor. Zero being not one completion, twenty-five being all have completed the mindfulness session.
Participant feedback via Questionnaire on the usefulness of the mindfulness experience on their emotional management and decision making process. | 1 year
  Two sets of questions asking about level of satisfaction with the mindfulness experience and how it pertains to their treatment decision satisfaction with responses being; 1. Not at all, 2. A little bit, 3. Somewhat, 4. Quite a bit, 5. Very much;
Feasibility of a mindfulness intervention prior to the surgical consultation by a single question regarding mode of communication participants prefer. | 1 year
  Options include by phone, video conference, or in-person
Feasibility of a mindfulness intervention prior to the surgical consultation by calculating proportion of participants who consent to the study. | 1 year
  Measurement will be done by looking at the ratio of participants approached versus participants consented to the study.
Feasibility of a mindfulness intervention prior to the surgical consultation by proportion of participants who have contact with the mindfulness teacher. | 1 year
  Measurement will be done by looking at the ratio of participants consented versus participants completed the mindfulness intervention with the teacher.
Feasibility of a mindfulness intervention prior to the surgical consultation by measuring the length of time to schedule the participant with the mindfulness teacher. | 1 year
  This will be measured by comparing date the participant consented on the study to the date participant had successfully scheduled their mindfulness session.
Feasibility of a mindfulness intervention prior to the surgical consultation by adherence to the mindfulness excercises. | 1 year
  The mindfulness instructor will conduct a follow-up session with the participant following their surgical consultation and measure the number of times the participant listened to the audio recordings given to them following their mindfulness session but prior to their surgical consultation.

SECONDARY OUTCOMES:
Patient Reported Outcomes on anxiety | 2 years
  using the HOSPITAL ANXIETY AND DEPRESSION SCALE (HADS); multiple choice, 4 point range scale. Examples: a. Most of the time b. A lot of the time c. From time to time, occasionally d. Not at all
Patient Reported Outcomes on fear of recurrence | 2 years
  using the Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire. Scale ranging from 1-strongly disagree to 5-strongly agree. Example: Because cancer is unpredictable, I feel I cannot plan for the future. (1 -Strongly Disagree,2- Disagree,3- Not Certain,4- Agree 5-Strongly Agree)
Patient Reported Outcomes on quality of life | 2 years
  utilizing the LINEAR ANALOGUE SELF ASSESSMENT (LASA) scale; Scale ranging from 0-10 with 0-being as bad as it can be, and 10 being as good as it can be. Last question on anxiety is flipped, 0-being no anxiety, and 10-being anxiety is as bad as it can be.
Patient Reported Outcomes on decisional satisfaction | 2 years
  Using the Decisional satisfaction questionnaire. Scale ranges 1-4 with 1-being very dissatisfied, to 4-very satisfied. Example: With your breast area in mind, in the past 2 weeks, how satisfied or dissatisfied have you been with How you look in the mirror clothed? 1-very dissatisfied 2-somewhat dissatisfied 3-somewhat satisfied 4-very satisfied;
Patient Reported Outcomes on mindfulness outcome | 2 years
  using the Mindfulness outcome measures (MeditationHX) Scale Ranges from 1-5 (1-Not at all, 2-A little bit, 3-Somewhat, 4-Quite a bit, 5-Very much) Example: Overall, I am satisfied with my experience participating in this research program (1-Not at all, 2-A little bit, 3-Somewhat, 4-Quite a bit, 5-Very much)
Patient Reported Outcomes and value concordant decision making | 2 years
  ratio measured by a formula used in previous studies

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Yao, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yao K, Belkora J, Bedrosian I, Rosenberg S, Sisco M, Barrera E, Kyrillios A, Tilburt J, Wang C, Rabbitt S, Pesce C, Simovic S, Winchester DJ, Sepucha K. Impact of an In-visit Decision Aid on Patient Knowledge about Contralateral Prophylactic Mastectomy: A Pilot Study. Ann Surg Oncol. 2017 Jan;24(1):91-99. doi: 10.1245/s10434-016-5556-x. Epub 2016 Sep 21. PMID 27654108
- [Background] Sepucha K, Ozanne E, Silvia K, Partridge A, Mulley AG Jr. An approach to measuring the quality of breast cancer decisions. Patient Educ Couns. 2007 Feb;65(2):261-9. doi: 10.1016/j.pec.2006.08.007. Epub 2006 Oct 4. PMID 17023138
- See also: Full Catastrophe Living: Using the Wisdom of your Mind to Face Stress, Pain and Illness. — https://www.scirp.org/reference/ReferencesPapers.aspx?ReferenceID=888540